CLINICAL TRIAL: NCT03426891
Title: A Phase I Trial of Pembrolizumab and Vorinostat Combined With Temozolomide and Radiation Therapy for Newly Diagnosed Glioblastoma
Brief Title: Pembrolizumab and Vorinostat Combined With Temozolomide for Newly Diagnosed Glioblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC-19342
Record Dates: First submitted 2018-02-02; First posted 2018-02-08 (Actual); Results first posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Glioblastoma; Brain Tumor; GBM
Keywords: Immunotherapy; Radiotherapy; Glioblastoma
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — pembrolizumab; Immunotherapy; Vorinostat; Drug Therapy; Histone Deacetylase Inhibitors; Temozolomide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose Escalation Phase (Experimental): Level -1: Vorinostat 100 mg/day PO during RTX; 300 mg/day PO after RTX Level 1: Vorinostat 200 mg/day PO during RTX; 300 mg/day PO after RTX
  Interventions: Drug: Pembrolizumab; Drug: Vorinostat; Drug: Temozolomide; Radiation: Radiotherapy
- Radiotherapy and Maintenance Phase (Experimental): 100 mg/day Vorinostat (+200 mg Pembro) with radiotherapy and 400 mg/day Vorinostat (+200 mg Pembro) maintenance.
  Interventions: Drug: Pembrolizumab; Drug: Vorinostat; Drug: Temozolomide; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Pembrolizumab — 200 mg intravenously (IV) every 3 weeks. The dose of pembrolizumab will remain the same throughout study treatment. During the maintenance phase, participants will receive pembrolizumab (for 12 months).
  Other Names: Keytruda; immunotherapy
Drug: Vorinostat — Dose Escalation Level -1 vorinostat 100 mg/day by mouth on days 1-5 every week during radiotherapy starting on first day of radiotherapy and 300 mg/day 1 week on 1 week off after radiotherapy. Level 1:vorinostat 200 mg/day by mouth on day 1-5 every week during radiotherapy, starting on first day of radiotherapy; and 300 mg/day 1 week on 1 week off after radiotherapy. Dose Escalation Level 2: vorinostat 300 mg/day by mouth on days 1-5 every week during radiotherapy, starting on first day of radiotherapy; and 400 mg/day 1 week on 1 week off after radiotherapy.
  Other Names: Zolinza™; chemotherapy; histone deacetylase inhibitor
Drug: Temozolomide — All participants will receive standard Temozolomide: Temozolomide (chemotherapy) 75 mg/m^2/day by mouth administered during the course of radiotherapy. Temozolomide will be administered continuously from Day 1 of radiotherapy to the last day of radiation. Maintenance Phase: temozolomide will start 4 weeks (+/- 3 days) after last dose of radiotherapy and will continue for 6 cycles post radiotherapy (150-200 mg/m^2/day, days 1-5 every 4 weeks) as per standard of care. During the maintenance phase, participants will receive Temozolomide (for the first 6 months).
  Other Names: chemotherapy; Temodar; TMZ
Radiation: Radiotherapy — All participants will receive standard radiotherapy: a total dose of 60 Gy administered in daily doses of 2 Gy, typically on a 5 days on / 2 days off schedule over 6 - 7 weeks.
  Other Names: radiation therapy

SUMMARY:
The purpose of this research study is to test the safety and tolerability of the combination treatment of the investigational drugs vorinostat and pembrolizumab, in combination with chemotherapy (temozolomide), and radiotherapy. The U.S. Food and Drug Administration (FDA) has approved pembrolizumab for use to treat a deadly skin cancer called melanoma and lung cancer and vorinostat to treat some forms of blood and lymph node cancers. However, both vorinostat and pembrolizumab are considered investigational drugs in this study because they are not approved for treatment of glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed glioblastoma or gliosarcoma
* Histologically confirmed diagnosis of World Health Organization Grade IV malignant glioma
* An interval of ≥ 21 days since surgical resection prior to treatment on the trial
* Karnofsky performance status of 70 or higher
* Adequate organ function laboratory values
* Resting baseline O2 saturation by pulse oximetry of ≥ 92% at rest
* Willing and able to provide written informed consent/assent for the trial.
* Life expectancy ≥ 12 weeks
* Willingness to discontinue medications known to be associated with risk of Torsades de Pointes such as quinidine, procainamide, disopyramide, amiodarone, erythromycin, clarithromycin, chlorpromazine and haloperidol
* Single lesion < 4 cm in longest diameter (diameter of enhancing lesion)
* Patient shouldn't have received any anti-cancer therapy for glioblastoma in past
* Females of childbearing potential (FOCBP) should have a negative urine or serum pregnancy prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Females and males of childbearing potential must be willing to use an adequate method of contraception per protocol for the course of the study through 120 days after the last dose of study medication. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for participant.
* Use of Optune device is allowed.

Exclusion Criteria:

* Had prior treatment of glioblastoma (GBM) with radiation and temozolomide
* Has evidence of leptomeningeal disease
* Had prior treatment with Gliadel
* Unable (due to existent medical condition) or unwilling to have a contrast enhanced MRI of brain
* Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. Physiologic doses of steroid therapy (≤ 2 mg/day dexamethasone equivalents) by the time of first dose of treatment are allowed.
* Has a known history of active Bacillus Tuberculosis (TB)
* Hypersensitivity to pembrolizumab or any of its excipients
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent. Note: Potential participants with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study. Note: If patient received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Patients with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Patients that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Patients with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study.
* Has known history of, or any evidence of active, interstitial lung disease or non-infectious pneumonitis requiring corticosteroid therapy
* Has an active serious infection requiring systemic therapy
* Had major surgical procedure, open biopsy, or significant traumatic injury within 21 days prior to day 1 of treatment on study
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2021-10-18 (Actual); Study Completion 2023-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Forsyth, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/

RESULTS

PARTICIPANT FLOW:
Groups:
- Level -1: Level -1: Vorinostat 100 mg/day PO during RTX; 300 mg/day PO after RTX
- Level 1: Level 1: Vorinostat 200 mg/day PO during RTX; 300 mg/day PO after RTX
Period: Overall Study
Arm/Group | Level -1 | Level 1 | Radiotherapy and Maintenance Phase
Started | 6 | 8 | 7
Completed | 6 | 8 | 6
Not Completed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Multiple dose levels are specified in the protocol but only the administered doses are included in the baseline characteristics.
Groups:
- Total: Total of all reporting groups
Arm/Group | Level -1 | Level 1 | Radiotherapy and Maintenance Phase | Total
Number analyzed (Participants) | 6 | 8 | 7 | 21
Age, Continuous [Mean (Full Range); unit: years] | 56.33 [36 to 67] | 60.38 [44 to 74] | 55.57 [32 to 77] | 57.62 [32 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 1 | 8
  Male | 4 | 3 | 6 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 2
  Not Hispanic or Latino | 5 | 7 | 5 | 17
  Unknown or Not Reported | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 5 | 7 | 5 | 17
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 6 | 8 | 7 | 21

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The maximum tolerated dose (MTD)/recommended dose expansion dose of vorinostat given in combination with pembrolizumab, temozolomide, and radiotherapy in patients with newly diagnosed glioblastoma. Toxicities will be graded in severity according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 for toxicity categories as outlined in the study protocol.
Time Frame: 12 weeks
Measure: Number; unit: mg/day Vorinostat
Arm/Group | Dose Escalation Phase
Number analyzed (Participants) | 14
mg/day Vorinostat
  MTD during RTX | 100
  MTD after RTX | 300

2. Secondary Outcome: Overall Survival (OS)
Description: Median overall survival rate, 95% confidence survival. OS: Time from randomization until death from any cause.
Time Frame: Up to 24 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Level -1 | Level 1 | Radiotherapy and Maintenance Phase
Number analyzed (Participants) | 6 | 8 | 7
Months | NA [17.9 to NA] — Follow-up period is too short to estimate | 12.2 [10.7 to NA] — Follow-up period is too short to estimate | NA [16.2 to NA] — Follow-up period is too short to estimate

ADVERSE EVENTS:
Time Frame: 2 years
Description: Adverse events were collected in aggregate at each dose level and were not captured per intervention.
Arm/Group | Level -1 | Level 1 | Radiotherapy and Maintenance Phase
All-Cause Mortality (participants affected / at risk) | 3/6 | 5/8 | 1/7
Serious Adverse Events (participants affected / at risk) | 2/6 | 6/8 | 3/7
Other Adverse Events (participants affected / at risk) | 6/6 | 8/8 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Level -1 (N=6) | Level 1 (N=8) | Radiotherapy and Maintenance Phase (N=7)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0)
Flu like symptoms (General disorders) | 1 (1) | 0 (0) | 0 (0)
Localized edema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Mania (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 1 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Level -1 (N=6) | Level 1 (N=8) | Radiotherapy and Maintenance Phase (N=7)
Lymphocyte count decreased (Investigations) | 6 (31) | 6 (17) | 6 (42)
Platelet count decreased (Investigations) | 6 (17) | 6 (15) | 6 (18)
Investigations - Other, specify (Investigations) | 5 (18) | 0 (0) | 7 (20)
White blood cell decreased (Investigations) | 3 (5) | 3 (4) | 4 (17)
Alanine aminotransferase increased (Investigations) | 3 (12) | 4 (14) | 2 (7)
Aspartate aminotransferase increased (Investigations) | 3 (6) | 4 (7) | 2 (5)
Creatinine increased (Investigations) | 2 (2) | 1 (3) | 4 (6)
Neutrophil count decreased (Investigations) | 2 (4) | 2 (3) | 2 (3)
Weight loss (Investigations) | 1 (2) | 2 (3) | 2 (4)
Alkaline phosphatase increased (Investigations) | 1 (1) | 2 (3) | 1 (1)
Lipase increased (Investigations) | 1 (4) | 0 (0) | 1 (1)
Weight gain (Investigations) | 1 (1) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (2)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Serum amylase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 5 (8) | 5 (6) | 4 (5)
Fever (General disorders) | 0 (0) | 2 (3) | 3 (4)
Localized edema (General disorders) | 2 (2) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 2 (2) | 0 (0) | 0 (0)
Irritability (General disorders) | 1 (1) | 0 (0) | 1 (1)
Edema face (General disorders) | 0 (0) | 1 (1) | 0 (0)
Facial pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Flu like symptoms (General disorders) | 1 (1) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 3 (5) | 1 (1) | 2 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 2 (4)
Hypermagnesemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 2 (4) | 3 (4) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 2 (3)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 3 (5) | 2 (5)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (12)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (2)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 5 (9) | 4 (8) | 6 (14)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (4)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 3 (3) | 1 (1)
Dysphasia (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3)
Dysgeusia (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (2) | 2 (2)
Seizure (Nervous system disorders) | 1 (2) | 2 (2) | 0 (0)
Tremor (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Edema cerebral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus pain (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (8) | 2 (2) | 4 (7)
Vomiting (Gastrointestinal disorders) | 5 (9) | 2 (2) | 3 (6)
Diarrhea (Gastrointestinal disorders) | 4 (8) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (4) | 0 (0) | 0 (0)
Fecal incontinence (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (6) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (5) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (3)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 3 (3) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 3 (3) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (2)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0)
Delusions (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Mania (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Psychosis (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 4 (4) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (3)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 1 (3)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (2)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (3) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (3) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Flashing lights (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Floaters (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 2 (2) | 0 (0)
Immune system disorders - Other, specify (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Vaginal inflammation (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-05): https://cdn.clinicaltrials.gov/large-docs/91/NCT03426891/Prot_SAP_000.pdf